CLINICAL TRIAL: NCT02976662
Title: Removal of Blastocoel Fluid Before Blastocyst Vitrification by Laser Pulse and Its Effect on Clinical Outcomes
Brief Title: Artificial Shrinkage for Human Blastocyst Prior Vitrification
Acronym: AS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dar AlMaraa Center (Other)
Collaborators: Benha University (Other)
Responsible Party: Principal Investigator, Yasmin, Scientific IVF lab director, Dar AlMaraa Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 006735
Record Dates: First submitted 2016-11-25; First posted 2016-11-29 (Estimated); Last update posted 2016-11-29 (Estimated); Status verified 2016-11

CONDITIONS: Vitrification

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Artificial shrinkage (Experimental): Elimination of blastocoelic fluid by creating a large hole in the zona pellucida at the cellular junction of the trophectoderm cells located far away from the inner cell mass with a laser pulse before vitrification.
  Interventions: Procedure: Artificial shrinkage
- Without Artificial shrinkage (No Intervention): Vitrify expanded blastocysts.

INTERVENTIONS:
Procedure: Artificial shrinkage — Artificially eliminated blastocoelic fluid before vitrification procedures.
  Arms: Artificial shrinkage

SUMMARY:
Investigators aim to investigate the effect of elimination of blastocoelic fluid by creating a large hole in the zona pellucida at the cellular junction of the trophectoderm cells located far away from the inner cell mass with a laser pulse before vitrification.

DETAILED DESCRIPTION:
Human blastocyst formation begins about 5 days after injecting a single sperm into an oocyte in ICSI cycle or incubation of them in IVF cycle. Human blastocyst consists of cells forming an outer layer called trophotoderm that will form the placenta in case of successful implantation, an inner cell mass which become the fetus, a fluid-filled blastocoel cavity in the center, and a surrounding zone pellucida from which the embryo hatches to implant in the uterus. Human blastocyst contains a large amount of liquid in the blastocoel, which alters the infiltration of vitrification solution during the vitrification procedures leading to ice crystal formation. Therefore, investigators need to compare blastocyst survival, clinical pregnancy and implantation rates between vitrified untreated expanded blastocysts and vitrified blastocysts with artificially eliminated blastocoels by a laser pulse prior to vitrification

ELIGIBILITY:
Inclusion Criteria:

* BMI of ≤ 32

Exclusion Criteria:

* Non-expanded blastocysts.
* Women who had uterine pathology or abnormality.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Implantation rate | 1 month
  number of intrauterine gestational sacs over the total number of embryos transferred

CONTACTS AND LOCATIONS:
Locations (1):
- Yasmin Magdi, Banhā, Egypt